CLINICAL TRIAL: NCT07261462
Title: The Effects of a Short-Term Isometric Exercise Program Targeting Tongue, Jaw, and Trunk Muscles on Muscle Strength and Synergistic Relationships in Post-Stroke Patients: A Single-Group Pre-Post Study
Brief Title: Oropharyngeal and Trunk Muscle Interactions After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, Assist Prof., Necmettin Erbakan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUPT202502; Necmettin Erbakan University (Other: Necmettin Erbakan University)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Back muscles; Post-stroke; Tongue strength; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All participants included in the study provided informed voluntary consent. The study was conducted in a single-blind manner, with the researcher who performed the patient assessments being different from the specialist who administered the exercise intervention. Inclusion criteria were: being within the first 30 days of stroke onset; being between 18 and 80 years of age; having experienced their first stroke; undergoing inpatient physical therapy and rehabilitation; and voluntarily consenting to participate. Exclusion criteria were: cognitive impairment, severe aphasia or communication difficulties, a history of other neurological diseases, a history of surgery in the oral or jaw region, and refusal to participate.
Masking Description: The study was conducted with a single group, and all participants received the exercise intervention. Assessments were performed by the researcher, and no blinding was applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Program (Experimental): All participants received isometric strengthening exercises twice daily for 14 days, with each session lasting approximately 30-40 minutes. Each exercise was performed for 15 repetitions, with each repetition held for 5 seconds followed by a rest. The exercise program included the following:
  Isometric Exercises for Tongue Muscles: Using a tongue depressor, patients were instructed to press their tongue forward, upward, downward, and to the sides against the depressor. These exercises aim to increase the strength of the tongue muscles, which play a critical role in swallowing function.
  Isometric Exercises for Jaw Muscles: Patients were asked to perform a chin tuck while in a supine position by tucking their chin toward their chest. Additionally, they were asked to place a soft ball under their chin and press against it to create an isometric contraction. These exercises target the muscles that facilitate swallowing.
  Isometric Exercises for Back Muscles: Patients who could not
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Isometric Exercises for Tongue Muscles: Using a tongue depressor, patients were instructed to press their tongue forward, upward, downward, and to the sides against the depressor. These exercises aim to increase the strength of the tongue muscles, which play a critical role in swallowing function .
  Isometric Exercises for Jaw Muscles: Patients were asked to perform a chin tuck while in a supine position by tucking their chin toward their chest. Additionally, they were asked to place a soft ball under their chin and press against it to create an isometric contraction. These exercises target the muscles that facilitate swallowing.
  Isometric Exercises for Back Muscles: Patients who could not sit with proper balance performed the exercises in a supine position with a soft ball placed under their back. They were asked to press their back against the ball to perform an isometric contraction. Patients with sufficient sitting balance were instructed to sit upright, pressing their backs

SUMMARY:
Background:This study aimed to investigate the effects of a short-term tongue-jaw-back isometric exercise program on these muscle groups and their interrelationships in the post-stroke period.

Methods: Twelve post-stroke patients were included in the study. A 14-day exercise program, consisting of two daily sessions targeting the tongue, jaw, and back muscles, was administered. Anterior and posterior tongue muscles, jaw muscles, and back muscle strength were assessed before and after the exercise program. Tongue pressure was measured using the Iowa Oral Performance Instrument (IOPI), chewing strength with a hand-held dynamometer, and back strength with a stabilizing pressure biofeedback unit.

Results: After the 14-day isometric exercise program, anterior tongue strength (p = 0.025), posterior tongue strength (p = 0.021), and back muscle strength (p = 0.005) showed significant increases compared to pre-treatment values. No significant change was observed in jaw strength (p = 0.475). Spearman correlation analysis revealed no significant relationships between tongue muscles and jaw or back muscles before treatment, and simple correlations after treatment also did not reach significance. However, partial correlation analysis showed that the relationship between tongue muscles was significantly influenced by jaw strength (p = 0.040) and back strength (p = 0.038) after the intervention.

Conclusions: Short-term isometric exercises targeting tongue, jaw, and back muscles in post-stroke patients effectively increased tongue and back muscle strength and enhanced the synergistic relationship among these muscle groups.

DETAILED DESCRIPTION:
Methods This study was designed as a single-group pre-post trial. A total of 12 post-stroke patients were included. All participants underwent a 14-day isometric exercise program targeting the tongue, jaw, and trunk muscles, with two daily sessions.

Study Design and Ethical Approval This study was designed as a prospective, single-center research project conducted at the Department of Physical Medicine and Rehabilitation, Meram Faculty of Medicine, Necmettin Erbakan University. Ethical approval for the study was obtained from the Necmettin Erbakan University Health Sciences Scientific Research Ethics Committee with decision number 2021/13-71. All participants included in the study provided informed voluntary consent. The study was conducted in a single-blind manner, with the researcher who performed the patient assessments being different from the specialist who administered the exercise intervention.

Participants Twelve patients with a diagnosis of acute ischemic or hemorrhagic stroke, who were hospitalized in the Physical Medicine and Rehabilitation service between February 2022 and December 2022, were enrolled in the study. Inclusion criteria were: being within the first 30 days of stroke onset; being between 18 and 80 years of age; having experienced their first stroke; undergoing inpatient physical therapy and rehabilitation; and voluntarily consenting to participate. Exclusion criteria were: cognitive impairment, severe aphasia or communication difficulties, a history of other neurological diseases, a history of surgery in the oral or jaw region, and refusal to participate.

Outcome Measures

The participants' sociodemographic data (age and stroke duration) were recorded. The following clinical and functional assessments were performed both before and after the 14-day program:

Motor Functional Status: Brunnstromm stages were used to evaluate motor recovery levels (upper extremity, hand, and lower extremity) of the hemiplegic side.

Functional Independence Status: The Barthel Index was used to determine the participants' level of independence in daily living activities.

Dysphagia Assessment: The Eating Assessment Tool-10 (EAT-10) score was used to determine the severity of swallowing difficulty.

Tongue Pressure Measurement: The Iowa Oral Performance Instrument (IOPI) was used to assess tongue muscle strength. For Anterior Tongue Pressure (ATP), the IOPI bulb was placed longitudinally along the hard palate, behind the alveolar ridge. For Posterior Tongue Pressure (PTP), the bulb was positioned at the posterior border of the hard palate. Both measurements were repeated three times, and the mean values were recorded.

Chewing Muscle Strength Measurement: Chewing muscle strength, representing masticatory force, was measured using a hand-held dynamometer. Participants were instructed to perform a jaw-opening movement against the dynamometer placed under the chin. This measurement was repeated three times, and the average value was used for analysis.

Back Muscle Strength Measurement: Back muscle strength was measured with a stabilizing pressure biofeedback unit. Individuals were asked to lie supine on a treatment table with their head turned to one side and knees flexed. These measurements were repeated three times, and the mean value was recorded.

Exercise Program

All participants received isometric strengthening exercises twice daily for 14 days, with each session lasting approximately 30-40 minutes. Each exercise was performed for 15 repetitions, with each repetition held for 5 seconds followed by a rest. The exercise program included the following:

Isometric Exercises for Tongue Muscles: Using a tongue depressor, patients were instructed to press their tongue forward, upward, downward, and to the sides against the depressor. These exercises aim to increase the strength of the tongue muscles, which play a critical role in swallowing function.

Isometric Exercises for Jaw Muscles: Patients were asked to perform a chin tuck while in a supine position by tucking their chin toward their chest. Additionally, they were asked to place a soft ball under their chin and press against it to create an isometric contraction. These exercises target the muscles that facilitate swallowing.

Isometric Exercises for Back Muscles: Patients who could not sit with proper balance performed the exercises in a supine position with a soft ball placed under their back. They were asked to press their back against the ball to perform an isometric contraction. Patients with sufficient sitting balance were instructed to sit upright, pressing their backs against a chair to engage their trunk muscles. Strengthening the trunk muscles in this manner supports overall postural control and swallowing stability.

ELIGIBILITY:
Inclusion Criteria:

* being within the first 30 days of stroke onset
* being between 18 and 80 years of age
* having experienced their first stroke
* undergoing inpatient physical therapy and rehabilitation
* voluntarily consenting to participate

Exclusion Criteria:

* cognitive impairment
* severe aphasia or communication difficulties
* a history of other neurological diseases
* a history of surgery in the oral or jaw region
* refusal to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Motor Functional Status | The following clinical and functional assessments were performed both before and after the 14-day program
  Brunnstromm stages were used to evaluate motor recovery levels (upper extremity, hand, and lower extremity) of the hemiplegic side

SECONDARY OUTCOMES:
Functional Independence Status | The following clinical and functional assessments were performed both before and after the 14-day program
  The Barthel Index was used to determine the participants' level of independence in daily living activities

OTHER OUTCOMES:
Dysphagia Assessment | The following clinical and functional assessments were performed both before and after the 14-day program
  The Eating Assessment Tool-10 (EAT-10) score was used to determine the severity of swallowing difficulty
Dysphagia Assessment | The following clinical and functional assessments were performed both before and after the 14-day program:
  The Eating Assessment Tool-10 (EAT-10) score was used to determine the severity of swallowing difficulty
Tongue Pressure Measurement | The following clinical and functional assessments were performed both before and after the 14-day program
  The Iowa Oral Performance Instrument (IOPI) was used to assess tongue muscle strength. For Anterior Tongue Pressure (ATP), the IOPI bulb was placed longitudinally along the hard palate, behind the alveolar ridge. For Posterior Tongue Pressure (PTP), the bulb was positioned at the posterior border of the hard palate. Both measurements were repeated three times, and the mean values were recorded.
Chewing Muscle Strength Measurement | The following clinical and functional assessments were performed both before and after the 14-day program
  Chewing muscle strength, representing masticatory force, was measured using a hand-held dynamometer. Participants were instructed to perform a jaw-opening movement against the dynamometer placed under the chin. This measurement was repeated three times, and the average value was used for analysis.
Back Muscle Strength Measurement | The following clinical and functional assessments were performed both before and after the 14-day program
  Back muscle strength was measured with a stabilizing pressure biofeedback unit. Individuals were asked to lie supine on a treatment table with their head turned to one side and knees flexed. These measurements were

CONTACTS AND LOCATIONS:
Locations (1):
- Nezahat Keleşoğlu Faculty of Health Sciences, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
ndividual participant data (IPD) will not be shared because of ethical and privacy restrictions.

REFERENCES:
- See also: Effects of Tongue-Strengthening Exercise on Tongue Strength Reserve and Detraining Effects among Healthy Adults: A Randomized Controlled Trial — https://pmc.ncbi.nlm.nih.gov/articles/PMC9180874/